CLINICAL TRIAL: NCT02077504
Title: Magnetoencephalographic Study of Glial Tumors Electromagnetic Signature
Brief Title: Glial Tumors Electromagnetic Signature Study by MagnetoEncephaloGraphy (MEG) "CONDUCTOME"
Acronym: CONDUCTOME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CONDUCTOME
Record Dates: First submitted 2013-09-18; First posted 2014-03-04 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Primitive Tumor With Chirurgical Indication
MeSH Terms: interventions — Magnetoencephalography; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CONDUCTOME (Experimental): MEG and MRI
  Interventions: Other: MEG and MRI

INTERVENTIONS:
Other: MEG and MRI — CONDUCTOME

SUMMARY:
The purpose of this study is to determine the correlation between functional MEG analysis of the tumor and its periphery and the tumor stage and treatment response.

DETAILED DESCRIPTION:
A better tumor grade definition would provide an optimized surgical care, prognosis and therapeutical response evaluation.

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old
* patient affiliated to social security or similarly regime
* informed consent form signed
* supra-tentorial primitive cerebral tumor

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Magnetic Resonance Imaging (MRI) contraindication (implanted material non MRI-compatible, ferro-magnetic foreign body, claustrophobia)
* Patients needed emergency medical care for other pathology
* severely altered general health (Performance Status 3 or 4)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-09; Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Magnetoencephalography (MEG) and Magnetic Resonance Imaging (MRI) data in tumor grade prediction | 1 week before exeresis
anatomopathologic and clinical data in tumor grade prediction | 1 week after exeresis

SECONDARY OUTCOMES:
Measurement of molecules involved in glial cells neuralisation expression in tumor samples | Up to 1 month after surgery
Tumoral growth modelisation from patient MEG and MRI data | Up to 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: François BERGER, MD, PhD, Principal Investigator — University Grenoble Hospital
Locations (1):
- CLINATEC, Grenoble, France